CLINICAL TRIAL: NCT00433849
Title: Switch and Maintenance Study of Subcutaneous or Intravenous Injections of R744 to Peritoneal Dialysis Patients (Phase Ⅲ Study)
Brief Title: Clinical Study of R744 to Peritoneal Dialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Chugai Pharmaceutical, Chugai Pharmaceutical
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JH20564
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Last update posted 2009-02-02 (Estimated); Status verified 2009-01

CONDITIONS: Peritoneal Dialysis Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: R744
- 2 (Experimental)
  Interventions: Drug: R744

INTERVENTIONS:
Drug: R744 — 100μg(i.v./p.o.)/4weeks for 8 weeks, then 25~400μg(i.v./p.o.)/4weeks for 40 weeks
  Arms: 1
Drug: R744 — 150μg(i.v./p.o.)/4weeks for 8 weeks, then 25~400μg(i.v./p.o.)/4weeks for 40 weeks
  Arms: 2

SUMMARY:
This study will assess the efficacy and safety of subcutaneous or intravenous R744 in renal anemia patients on Peritoneal Dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been receiving peritoneal dialysis for at least 12 weeks before registration
* Patients aged ≥ 20 years at the time of obtaining consent
* Patients who have been receiving a rHuEPO preparation at least once a month for at least 8 weeks before registration
* Patients whose mean value of Hb concentrations determined within 8 weeks before registration has been between 10.0 g/dL and <12.0 g/dL
* Patients whose transferrin saturation has been ≥ 20 % or ferritin has been ≥ 100ng/mL at any one time point within 8 weeks before registration

Exclusion Criteria:

* Patients with hardly controllable hypertension (patients whose diastolic blood pressure has been ≥ 100 mmHg on more than 1/3 of the determining occasions within 12 weeks before registration
* Patients with congestive cardiac failure (≥ Class III in NYHA cardiac function classification)
* Female patients who are pregnant, lactating, possibly pregnant or not willing to take a contraceptive measure in the period from the day of starting the treatment with the study drug to 90 days after the day of the last dose of the study drug
* Patients with complication of myocardial infarction, pulmonary infarction or cerebral infarction (excluding asymptomatic cerebral infarction)
* Patients confirmed to have serious allergy or serious drug allergy (shock, anaphylactoid symptom)
* Patients hypersensitive to a rHuEPO preparation
* Patients with malignant tumor (including hemic malignant tumor), severe infection, systemic hemic disease (osteomyelodysplasia syndrome, hemoglobinopathy, etc.), hemolytic anemia or apparent hemorrhagic lesion such as digestive tract hemorrhage
* Patients who have had an onset of peritonitis within 4 weeks before registration
* Patients who have received an anabolic hormone preparation, testosterone enanthate or mepitiostane within 12 weeks before registration
* Patients who have received another investigational drug within 12 weeks before registration
* Patients who have received R744 before registration
* Patients whose AST(GOT) value ≥ 100 IU/L or ALT(GPT) value ≥ 100 IU/L before registration
* Patients who have received erythrocyte transfusion within 16 weeks before registration
* Patients for whom a surgical operation accompanied by marked bleeding is planned during the study period
* In addition, patients who are judged as ineligible to participate in this study by the investigator or sub-investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-02; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Rate of patients who maintain Hb concentration in the range of ≥ 10.0g/dL and ≤ 12.0g/dL | 48 weeks

SECONDARY OUTCOMES:
Slope of regression line of Hb concentration (g/dL/week) | 48 weeks
Rate of patients who maintain Hb concentration in the range of baseline ± 1.0g/dL | 48 weeks
Rate of patients who maintain Hb concentration in the range of ≥ 10.0g/dL and < 13.0g/dL | 48 weeks
Laboratory measurements | 48 weeks
Adverse Event | 48 weeks
Anti-R744 antibody titer | 48 weeks
Vital signs, standard 12-lead ECG | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Takanori Baba, Study Chair — Clinical Research Department 2
Locations (6):
- Japan (6):
  - Chugoku/Shikoku region, Chugoku/Shikoku
  - Chubu region, Chūbu
  - Hokkaido/Tohoku region, Hokkaido/Tohoku
  - Kanto/Koshinetsu region, Kanto/Koshinetsu
  - Kinki/Hokuriku region, Kinki/Hokuriku
  - Kyusyu region, Kyusyu